CLINICAL TRIAL: NCT04745455
Title: An Open-label Single-arm Study to Investigate Gastrointestinal Tolerance, Safety, and Acceptability of a New Infant Formula Containing Prebiotics, Probiotics and Postbiotics, in Healthy Term Infants.
Brief Title: Gastrointestinal Tolerance and Safety of an Infant Formula Containing Prebiotics, Probiotics and Postbiotics.
Acronym: TREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SBB20R&32116
Record Dates: First submitted 2021-01-12; First posted 2021-02-09 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-01

CONDITIONS: Gastrointestinal Tolerance
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cow's milk based infant formula containing prebiotics, probiotics and postbiotics (Other)
  Interventions: Other: Infant formula containing prebiotics, probiotics and postbiotics

INTERVENTIONS:
Other: Infant formula containing prebiotics, probiotics and postbiotics — Infant formula containing prebiotics, probiotics and postbiotics

SUMMARY:
A study to investigate the gastrointestinal tolerance and safety of a new formula containing prebiotics, probiotics and postbiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Term infants with a gestational age at birth of ≥37 weeks + 0 days and ≤41 weeks + 6 days;
2. Singleton, healthy infants as judged by the principle investigator;
3. Infants with age at screening ≥2 weeks (14 days) and ≤ 12 weeks (84 days)
4. Infants who are fully formula fed for at least 1 week prior to screening and whose parents have autonomously decided to fully formula feed, i.e. not to breastfeed or have ended breastfeeding, and who are intending to fully formula feed;
5. Written informed consent from the parent(s) and/or legally acceptable representative(s), aged ≥ 18 years.

Exclusion Criteria:

1. Infants who require to be fed a special diet other than standard cow's milk-based infant formula;
2. Infants known to have or suspected to have cow's milk protein allergy, lactose intolerance, or galactosaemia including history of any other allergic manifestations or known allergy to any of the study product ingredients;
3. Infants with known or suspected congenital diseases or malformations which could interfere with the study or its outcome parameters, such as but not limited to: GI malformations, congenital metabolic disorders, severe congenital cardiac disorders, immunodeficiency or major surgery, as per the clinical judgment of the Investigator;
4. Infants diagnosed with a gastrointestinal infection within 4 weeks prior to screening;
5. Infants with current or previous illnesses/conditions or interventions which could interfere with the study or its outcome parameters (e.g. diarrhea requiring treatment, constipation requiring treatment, regurgitation requiring treatment, dental/medical procedures which may impact oral feeding), as per the clinical judgment of the Investigator;
6. Received any of the following products/medication prior to screening: systemic antibiotics, prokinetics, proton pump inhibitors, prebiotic supplements, probiotic supplements, complementary feeding/weaning within 4 weeks prior to screening;
7. Incapability of infants' parents to comply with study protocol as per the judgment of the Investigator (e.g. fluency in local language, access to laptop/smartphone devices and internet connection required for data collection);
8. Infants with previous, current or intended participation in any other clinical study involving investigational or marketed products concomitantly or prior to study.

   -

Ages: 14 Days to 84 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | Baseline
  A 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress.
Gastrointestinal tolerance | Day 7
  A 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress.
Gastrointestinal tolerance | Day 14
  A 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress.
Gastrointestinal tolerance | Day 21
  A 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress.
Gastrointestinal tolerance | Day 28
  A 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress.

SECONDARY OUTCOMES:
Stool consistency | Baseline
  Parent reported daily stool consistency using stool scales with categories 1; watery, 2; loose, 3; formed, 4; hard
Stool consistency | Day 7
  Parent reported daily stool consistency using stool scales with categories 1; watery, 2; loose, 3; formed, 4; hard
Stool consistency | Day 14
  Parent reported daily stool consistency using stool scales with categories 1; watery, 2; loose, 3; formed, 4; hard
Stool consistency | Day 21
  Parent reported daily stool consistency using stool scales with categories 1; watery, 2; loose, 3; formed, 4; hard
Stool consistency | Day 28
  Parent reported daily stool consistency using stool scales with categories 1; watery, 2; loose, 3; formed, 4; hard
Stool frequency | Baseline
  Parent reported daily number of stools
Stool frequency | Day 7
  Parent reported daily number of stools
Stool frequency | Day 14
  Parent reported daily number of stools
Stool frequency | Day 21
  Parent reported daily number of stools
Stool frequency | Day 28
  Parent reported daily number of stools
Incidence, frequency, and severity of (S)AEs, and relatedness to study product of (Serious) Adverse Events. | Through study completion, an average of one month
  (S)AE collection

OTHER OUTCOMES:
Well being questionnaire | Baseline
  A parent reported 3-item questionnaire with individual scores from 1-5 (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree)
Well being questionnaire | Day 28
  A parent reported 3-item questionnaire with individual scores from 1-5 (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree)
Study product appreciation questionnaire; | Day 7
  A parent reported evaluation of product characteristics with a categorical rating scale and open questions
Study product appreciation questionnaire; | Day 28
  A parent reported evaluation of product characteristics with a categorical rating scale and open questions

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Poliklinika Ginekologiczno-Poloznicza Sp. Z.O.O Sp.K, Bialystok
  - Izabela Tarczoń Przylądek Zdrowia Specjalistyczne Poradnie Medyczne, Krakow
  - NZLA Michalkowice Jarosz i partnerzy Spolka, Siemianowice Śląskie

IPD SHARING:
Plan to Share IPD: No